CLINICAL TRIAL: NCT04874298
Title: The Effect of Ginger and Peppermint on Postoperative Nausea and Vomiting in Patients After Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sona PASHAEI (Other)
Responsible Party: Sponsor-Investigator, Sona PASHAEI, Lecturer, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-8-1
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Nausea, Vomiting, Postoperative Nausea and Vomiting, Ginger, Peppermint, Thyroid surgery, Nursing
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — ginger extract; peppermint oil

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study to determine the effect of ginger and peppermint after thyroid surgery on postoperative nausea and vomiting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Arm 1 (Ginger Group) (Experimental): Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental group. In the postoperative period at the 2nd, 4th, 6th, 12th and 24th hours, the patient will use ginger oil as inhalation. The structure of the inhaler tube is explained. The back cover of the inhaler tube is opened and absorbent cotton swab is inserted into it. Cotton swab 1 ml of essential oil is added by dropping on it. The back cover of the inhaler tube is closed. It is waited for 10-15 minutes. The front cover of the inhaler tube is opened at the time intervals specified in the study procedure (at the 2nd, 4th, 6th, 12th and 24th hours after the operation, and the patient is allowed to smell essential oil from the tube. With the end of the sniffing process, the front cover of the tube is closed and the essential oil remains in the tube. The essential oil tubes to be applied will be prepared separately for each patient and that day.
  Interventions: Other: Ginger
- Intervention Arm 2 (Peppermint Group) (Experimental): Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental group. In the postoperative period at the 2nd, 4th, 6th, 12th and 24th hours, the patient will use Peppermint oil as inhalation. The structure of the inhaler tube is explained. The back cover of the inhaler tube is opened and absorbent cotton swab is inserted into it. Cotton swab 1 ml of essential oil is added by dropping on it. The back cover of the inhaler tube is closed. It is waited for 10-15 minutes. The front cover of the inhaler tube is opened at the time intervals specified in the study procedure (at the 2nd, 4th, 6th, 12th and 24th hours after the operation, and the patient is allowed to smell essential oil from the tube. With the end of the sniffing process, the front cover of the tube is closed and the essential oil remains in the tube. The essential oil tubes to be applied will be prepared separately for each patient and that day.
  Interventions: Other: Peppermint
- Control Arm (No Intervention): In the control group, no application will be made during and after the surgical intervention, and routine treatment and care will be applied.

INTERVENTIONS:
Other: Ginger — Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental group. In the postoperative period at the 2nd, 4th, 6th, 12th and 24th hours, the patient will use Ginger and Peppermint oil as inhalation. The structure of the inhaler tube is explained. The back cover of the inhaler tube is opened and absorbent cotton swab is inserted into it. Cotton swab 1 ml of essential oil is added by dropping on it. The back cover of the inhaler tube is closed. It is waited for 10-15 minutes. The front cover of the inhaler tube is opened at the time intervals specified in the study procedure (at the 2nd, 4th, 6th, 12th and 24th hours after the operation, and the patient is allowed to smell essential oil from the tube. With the end of the sniffing process, the front cover of the tube is closed and the essential oil remains in the tube. The essential oil tubes to be applied will be prepared separately for each patient and that day.
  Arms: Intervention Arm 1 (Ginger Group)
Other: Peppermint — Peppermint
  Arms: Intervention Arm 2 (Peppermint Group)

SUMMARY:
The study was planned as a randomized controlled experimental study to determine the effect of inhalation use of ginger and peppermint on postoperative nausea and vomiting in patients undergoing thyroidectomy surgery. After the approval of the ethics committee and institutional permission, 81 patients who applied to the general surgery clinic for thyroidectomy between 1 December 2020 and 1 December 2021 and met the inclusion criteria will be included in the study. Within the scope of the planned study, the sample size in the light of the reported academic studies was determined as effect size d = 0.40 (effect size), α = 0.05 (margin of error), 1-β = 0.90 (Power) and by using the G-power package program with the specified criteria. It was decided to recruit 81 people (27 people per 3 group). Block randomization method will be used to determine the experimental and control groups. In order for the groups to be distributed homogeneously, the order produced by a computer program (https://www.randomizer.org/) will be used. Randomization will be done by a biostatistician outside the researcher. Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups according to the randomization list. Before the operation, the patient will be visited and information will be given about the purpose, content and intervention to be applied. After obtaining verbal and written permission from the patients who accepted to participate in the study, the "Informed Consent" will be filled in the "Patient Identification form. On the day of surgery, "surgical intervention information will be filled in by the researcher. In the postoperative period at the 2nd, 4th, 6th, 12th and 24th hours, the patient will use ginger and peppermint oil as inhalation. At the end of the 24th hour, the application will be terminated. In the control group, no application will be made during and after the surgical intervention, and routine treatment and care will be applied. After admission to the clinic of the patients in the experimental and control groups, the severity of pain, nausea and vomiting, the number of nausea-vomiting at the 2nd, 6th, 12th and 24th hours, the name, dose, frequency and time of the antiemetic drugs used were determined by the researcher. At the end of the 24th hour, Rhodes Nausea Vomiting Index score will be evaluated by the researcher.

DETAILED DESCRIPTION:
The universe of the research; patients who are planned to undergo thyroid surgery between 1 December 2020 and 1 December 2021 in the general surgery clinic where the study will be conducted will comprise the patients who meet the inclusion criteria and agree to participate in the study. The research was planned as a randomized controlled experimental study. Block randomization method will be used to determine the experimental and control groups. In order for the groups to be distributed homogeneously, the order produced by a computer program (https://www.randomizer.org/) will be used. Randomization will be done by a biostatistician outside the researcher. Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups according to the randomization list. Research data will be collected in a hospital's general surgery ward between 1 December 2020 and 1 December 2021.

Independent variables of the research; age, gender, educational status, marital status, height, weight, habits and general health parameters were defined as independent variables. The dependent variables of the study are postoperative nausea-vomiting status (number and severity), pain severity (Visual Analog Scale-VAS), and Rhodes nausea-vomiting index score average.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are 18 years old or older,
2. According to the American Association of Anesthesiologists (ASA) classification; ASA score I and II,
3. Not known ginger and peppermint allergy,
4. Patients who are qualified to understand and answer questions in terms of cognitive capacity,
5. Patients without any psychiatric disorder,
6. Patients who agree to participate in the study will be included in the study.

Exclusion Criteria:

1. Under 18 years old,
2. Those with nutritional disorders,
3. Patients who require additional treatment to prevent nausea and vomiting, or patients using non-prescription anti-nausea and other complementary therapy,
4. Patients with peppermint and ginger allergy,
5. Those who have additional diseases (gastrointestinal system diseases, central nervous system tumors, vertigo etc.) that may affect the state of nausea and vomiting,
6. Not agreeing to participate in the research,
7. Those with respiratory diseases such as asthma, COPD, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain severity | Reported pain severity in the first 24 hours after surgery
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst pain
The number of postoperative nausea, vomiting and retching | Reported the number of nausea, vomiting and retching in the first 24 hours after surgery
  The number of nausea, vomiting
Postoperative nausea and vomiting severity | Reported nausea and vomiting severity in the first 24 hours after surgery
  Nausea and vomiting severity with Visual Assessment Scale (VAS) Score: 0-10; 0- None, 10- Agonizing
Use of antiemetics | In the first 24 hours after surgery
  The name, dose, frequency and time of the antiemetic drugs
Rhodes Nausea Vomiting Index score | At the end of the 24th hour after surgery
  Evaluation of Rhodes Nausea Vomiting Index score In order to score the scale, responses to items 1, 3, 6 and 7 are calculated in reverse order; For each answer, they are scored as 0: minimum, 4: most discomfort, and the score obtained from 8 items is added. It is expressed as 32 points, the highest possible value.

SECONDARY OUTCOMES:
Postoperative complications | End of surgery to hospital discharge 2-3 days
  Evaluation of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz E Ersoy, Prof.Dr, Principal Investigator — Bezmialem University; Nuray AKYUZ, Dr, Study Director — Istanbul University - Cerrahpasa; Sona PASHAEI, MSC, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- IU-Cerrahpaşa Florence Nightingale Faculty of Nursing Department of Surgical Nursing Abide-i Hürriyet street. 34381 Sisli - Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No